CLINICAL TRIAL: NCT01939210
Title: Influence of Meditation-Based Breathing Training on Target Motion Management and Distress During Radiation for Abdominal and Lung Malignancies
Brief Title: Meditation-Based Breathing Training in Improving Target Motion Management and Reducing Distress in Patients With Abdominal or Lung Cancer Undergoing Radiation Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funding to hire a dedicated study interventionist
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Alyson Moadel, Principal Investigator, Albert Einstein College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 09-12-392; NCI-2013-01127 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 09-068; 09-12-392 (Other: Albert Einstein College of Medicine); P30CA013330 (NIH)
Record Dates: First submitted 2013-09-06; First posted 2013-09-11 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Anxiety; Depression; Digestive System Neoplasm; Lung Neoplasm; Pain; Post-Traumatic Stress Disorder; Psychological Impact of Cancer
MeSH Terms: conditions — Anxiety Disorders; Depression; Digestive System Neoplasms; Lung Neoplasms; Pain; Stress Disorders, Post-Traumatic | interventions — Early Intervention, Educational; Educational Status; Methods; Meditation

ARMS (2):
- Arm I (breathing training sessions) (Experimental): Patients participate in 3 50-minute breathing training sessions, including a psycho-educational component and meditation-based breathing training, over 10 days. Patients then undergo 4D-CT on day 14 and undergo image-guided SBRT or standard radiation therapy 5 times a week for up to 5 fractions or 25 fractions, respectively.
  Interventions: Other: Educational Intervention; Other: Meditation Therapy; Other: Questionnaire Administration
- Arm II (control) (Active Comparator): Patients receive standard care over 10 days. Patients then undergo 4D-CT on day 14 and undergo image-guided SBRT or standard radiation therapy 5 times a week for up to 5 fractions or 25 fractions, respectively.
  Interventions: Other: Questionnaire Administration

INTERVENTIONS:
Other: Educational Intervention — Participate in breathing training sessions
  Other Names: Education for Intervention; Intervention, Educational
  Arms: Arm I (breathing training sessions)
Other: Meditation Therapy — Participate in breathing training sessions
  Other Names: Meditation
  Arms: Arm I (breathing training sessions)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized pilot clinical trial studies the effects of meditation-based breathing training on patients' control of their breathing patterns and breathing-related movement, as well as on their psychological distress and treatment experience during radiation therapy. Meditation-based breathing training may decrease breathing-related movement and the amount of stress by improving breathing patterns in patients with abdominal or lung cancer undergoing radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the influence of regular breathing cycles using breathing relaxation techniques on efficacy of the respiratory-gated treatment as measured by: (1) real-time position management (RPM) parameters; (2) end inspiration or expiration length; (3) changes in gate width.

SECONDARY OBJECTIVES:

I. To evaluate the effect of breathing relaxation techniques on: (1) psychosocial outcomes; (2) treatment compliance.

OUTLINE:

PHASE I: Patients and staff members complete structured interviews at baseline.

PHASE II: Patients are randomized to 1 of 2 arms.

ARM I: Patients participate in 3 50-minute breathing training sessions, including a psycho-educational component and meditation-based breathing training, over 10 days. Patients then undergo four dimensional computed tomography (4D-CT) on day 14 and undergo image-guided stereotactic body radiation therapy (SBRT) or standard radiation therapy 5 times a week for up to 5 fractions or 25 fractions, respectively.

ARM II: Patients receive standard care over 10 days. Patients then undergo 4D-CT on day 14 and undergo image-guided SBRT or standard radiation therapy 5 times a week for up to 5 fractions or 25 fractions, respectively.

After completion of study treatment, patients are followed up at 2 or 5 weeks.

ELIGIBILITY:
Inclusion Criteria:

* PHASE I - PATIENTS: All patients with abdominal tumors who have undergone at least 4 respiratory-gated radiotherapy treatments
* PHASE I - PATIENTS: Full comprehension of English language
* PHASE I - STAFF: All staff who have overseen the delivery of respiratory-gated radiotherapy for at least 6 months
* PHASE I - STAFF: Full comprehension of English language
* PHASE II: All patients with abdominal or lung tumors undergoing a respiratory gating simulation
* PHASE II: Karnofsky performance status > 60%
* PHASE II: Life expectancy > 3 months
* PHASE II: No prior radiotherapy to the abdomen/lung
* PHASE II: Full comprehension of English language

Exclusion Criteria:

* PHASE I - PATIENTS: Inability to comprehend English language interview questions
* PHASE I - STAFF: Inability to comprehend English language interview questions
* PHASE II: Karnofsky performance status < 60%
* PHASE II: Prior radiotherapy to the abdomen/lung
* PHASE II: Evidence of progressive or untreated gross disease outside of the abdomen/lung
* PHASE II: Inability to comprehend English language breathing exercise instructions
* PHASE II: Concurrent diagnosis of a significant respiratory disorder which requires the use of oxygen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-02; Primary Completion 2015-06 (Actual); Study Completion 2015-12-02 (Actual)

PRIMARY OUTCOMES:
Change in duty cycle, defined as the fraction of the time of the breathing cycle that the beam is on, before and after breath coaching | Baseline to up to 5 weeks
  Data will be analyzed using a mixed-model analysis of variance (ANOVA) to test for differences between the two independent groups (with a fixed effect factor of group membership).
Changes in gate width | Baseline to up to 5 weeks
Changes in the length of the end expiration or end inspiration defined as when the breathing trace or internal motion change direction | Baseline to up to 5 weeks
  Data will be analyzed using a mixed-model ANOVA to test for differences between the two independent groups (with a fixed effect factor of group membership).

SECONDARY OUTCOMES:
Change in patients' self-reported levels of psychological distress, physical pain and discomfort, and post-traumatic stress associated with cancer diagnosis and radiation treatment | Baseline to up to 5 weeks
  Data will be analyzed using a mixed-model ANOVA to test for differences between the two independent groups (with a fixed effect factor of group membership).

CONTACTS AND LOCATIONS:
Overall Officials: Alyson Moadel, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States